CLINICAL TRIAL: NCT03096158
Title: Cardiac and Endothelial Function Response to Early Exercise Training (CEFREET Study) After Coronary Artery Bypass Surgery: a Randomized Clinical Trial
Brief Title: Cardiac and Endothelial Function Response to Early Exercise Training After Coronary Artery Bypass Surgery
Acronym: CEFREET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEFREET
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Bypass Grafting; Coronary Artery Disease; Cardiac Rehabilitation
Keywords: Coronary artery bypass grafting; Cardiorespiratory rehabilitation; Functional electrical stimulation; Inspiratory muscle training; Aerobic training; Isometric handgrip training; Functional capacity; Endothelial function; Cardiac function
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ventilatory Muscle Training (TREMVEN) (Experimental): The enrolled participants will perform inspiratory muscle training (IMT) for 20 minutes during the period of hospitalization, using the Power Breathe device (POWERbreathe International LTD). During training, subjects will be instructed to maintain diaphragmatic breathing at a rate at 15 to 20 breaths/min. The inspiratory load will be set at 30% of maximal static inspiratory pressure (PImax). It will be occur once per day until the hospital exit.
  Interventions: Other: Ventilatory Muscle Training (TREMVEN)
- Aerobic Training (AERO) (Experimental): It will consist of supervised walking, lasting 20 minutes a day, during the period of hospitalization of the participants. Heart rate (HR) will be constantly monitored through a cardiac monitor (Polar), with the objective of maintaining between 50 and 60% of the maximum HR predicted by age; Similar to 40 to 50% of VO2max. Blood pressure, oxygen saturation (SpO2) and level of dyspnea (Borg's effort perception scale) will also be monitored constantly. It will be occur once per day until the hospital exit.
  Interventions: Other: Aerobic Training (AERO)
- Isometric Handgrip Training (ISO) (Experimental): Study participants will perform 5 x 2 min alternating bilateral contractions of the hand flexor muscles at 30% maximum voluntary contraction with one minute rest between contractions, in a total of 20 minutes training during the period of hospitalization. It will be occur once per day until the hospital exit.
  Interventions: Other: Isometric Handgrip Training (ISO)

INTERVENTIONS:
Other: Ventilatory Muscle Training (TREMVEN) — Early cardiac rehabilitation after coronary artery bypass graft:
  The enrolled participants will perform IMT or P-IMT for 20 minutes during the period of hospitalization, using the Power Breathe device (POWERbreathe International LTD). During training, subjects will be instructed to maintain diaphragmatic breathing at a rate at 15 to 20 breaths/min. The inspiratory load will be set at 30% of maximal static inspiratory pressure (PImax). It will be occur once per day until the hospital exit.
  Arms: Ventilatory Muscle Training (TREMVEN)
Other: Aerobic Training (AERO) — Early cardiac rehabilitation after coronary artery bypass graft:
  It will consist of supervised walking, lasting 20 minutes a day, during the period of hospitalization of the participants. Heart rate (HR) will be constantly monitored through a cardiac monitor (Polar), with the objective of maintaining between 50 and 60% of the maximum HR predicted by age; Similar to 40 to 50% of VO2max. Blood pressure, SpO2 and level of dyspnea (Borg's effort perception scale) will also be monitored constantly. It will be occur once per day until the hospital exit.
  Arms: Aerobic Training (AERO)
Other: Isometric Handgrip Training (ISO) — Early cardiac rehabilitation after coronary artery bypass graft:
  Study participants will perform 5 x 2 min alternating bilateral contractions of the hand flexor muscles at 30% maximum voluntary contraction with one minute rest between contractions, in a total of 20 minutes training during the period of hospitalization. It will be occur once per day until the hospital exit.
  Arms: Isometric Handgrip Training (ISO)

SUMMARY:
Background: Coronary artery bypass grafting (CABG) due to coronary artery disease (CAD) is one of the main surgical procedures performed in the area of cardiology. Individuals undergoing CABG present sarcopenia, decreased muscle strength of the lower limbs, decreased respiratory muscle strength and dyspnea due to immobility in the bed and the inherent conditions of the disease itself. Cardiorespiratory rehabilitation techniques are rarely used with measurement in hospitals and can greatly favor an early and effective reestablishment to this population in several parameters. Objective: To evaluate the effect of functional electrical stimulation (FES), ventilatory muscle training (TREMVEN), early aerobic training (AERO) and isometric handgrip training (ISO) on the functional capacity, endothelial function and cardiac parameters of individuals undergoing CABG. Methods: In a randomized clinical trial, volunteers will be allocated into four groups: EEF, TREMVEN, AERO or ISO in the preoperative period of CABG. After 48 hours (postoperative midway) of the surgery, the protocol will begin until after hospital discharge. The endpoints evaluated will be: functional capacity, respiratory muscle strength, systolic and diastolic function, arterial endothelial function, inflammatory profile and plasma levels of vascular endothelial growth factor (VEGF). Scientific contributions: Phase 1 cardiorespiratory rehabilitation with alternative interventions may provide an increase in functional capacity, strengthening of respiratory muscles, improvement in cardiac and endothelial functions, as well as increased systemic VEGF levels (myocardial revascularization) and improvement of the inflammatory profile, effectively forwarding the individuals to the rehabilitation phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Be elective for the first CABG due to a previous ischemic event;
* Do not present other associated heart diseases;
* Absence of history of neuromuscular, autoimmune and infectious diseases;
* Age between 50 to 75 years;
* Signature of the Informed Consent Term.
* No hyperreactivity during the pre-intervention evaluation tests;
* No chronic renal failure; history of malignant disease with life expectancy <2 years;
* No severe arrhythmias, angina pectoris, pulmonary embolism and thrombophlebitis;
* Do not have orthopedic limitations or any physical or mental limitation that prevents the proposed exercises from being performed;
* Present Left Ventricular Ejection Fraction (LVEF) > 40% in 48h after CABG, and
* After the physical training period, individuals who have not completed a minimum of 80% of the protocol will be excluded from the sample due to refusal or withdrawal.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Functional Capacity - Six-Minute Walk Test (6MWT) | Pre and post (7 days) coronary artery bypass surgery
  The 6MWT will be performed to assess functional capacity following the guidelines proposed by the American Thoracic Society.

SECONDARY OUTCOMES:
Cardiac Function - Echocardiography | Pre and post (7 days) coronary artery bypass surgery
  A high resolution ultrasound device equipped with a 2-5 megahertz (MHz) transducer will be used to obtain two-dimensional echocardiographic parameters: left ventricular end-diastolic volume, left ventricular end-systolic volume, left ventricular ejection fraction (cardiac function). The images will be stored on the hard disk of the echocardiographic device and analyzed offline in specific software of the equipment itself.
Endothelial Function- Flow-Mediated Dilation (FMD) | Pre and post (7 days) coronary artery bypass surgery
  To examine brachial artery FMD, the arm will be extended and positioned at an angle of ~80° from the torso. A rapid inflation and deflation pneumatic cuff will be positioned on the forearm to provide an ischemia. A 10-MHz multi-frequency linear array probes, attached to a high resolution ultrasound machine, will be then used to image the brachial artery in the distal 1⁄3rd of the upper arm. Following baseline assessments, the forearm cuff will be inflated ( > 200 mmHg) for 5 minutes. Diameter and flow recordings resumed 30s prior to cuff deflation and continued for 3 minutes.
Femoral Quadriceps Perimetry | Pre and post (7 days) coronary artery bypass surgery
  Quadriceps perimetry will be measured every 5 cm, starting from the top edge of the patella in the proximal direction. Thus, measurements of 5, 10, 15 and 20 cm will be performed in both lower limbs.
Maximal Inspiratory Pressure | Pre and post (7 days) coronary artery bypass surgery
  Inspiratory muscle function testing will be performed using a pressure transducer (MVD-300), connected to a system with two unidirectional valves. PImax will be determined in deep inspiration from residual volume against an occluded airway with a minor air leak (2 mm). The highest pressure of six measurements (with less than 5% difference) will be used to define PImax.
Handgrip Strength | Pre and post (7 days) coronary artery bypass surgery
  A digital handgrip device will be held while sitting upright in a chair with feet flat on the floor and 5 maximal contractions of the hand flexor muscles with each hand will be performed to determine maximum voluntary contraction (MVC). 30% of MVC will be used to isometric handgrip resistance exercise.
ELISA Immunoassay | Pre and post (7 days) coronary artery bypass surgery
  A venous blood sample will be collected pre- and post-intervention. After centrifugation at 1.000 rpm for 10 min at 4 C, the plasma will be separated and stored at 80 C until assay. VEGF and inflammatory markers will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Bruna Eibel, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670